CLINICAL TRIAL: NCT02479529
Title: Weaning of Norepinephrine Guided by the Dynamic Arterial Compliance in Cardiac Surgery Post Operative.
Acronym: SNEAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2014_843_0014; 2014-002707-22 (EudraCT Number)
Record Dates: First submitted 2015-03-18; First posted 2015-06-24 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Vasoplegic Syndrome
MeSH Terms: conditions — Vasoplegia | interventions — Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- administration of norepinephrine by dynamic elastance (Experimental): The norepinephrine weaning strategy is based on an index that reflects the vasomotor tone: dynamic arterial elastance
  Interventions: Drug: Norepinephrine
- control administration of norepinephrine (Other): The usual procedure of withdrawal norepinephrine is based on hemodynamic parameters (blood pressure), clinical (cutaneous perfusion, mottling, hourly diuresis) and biological (SVO2, arterial lactate).
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — Administration and weaning of norepinephrine is based on dynamic arterial elastance
  Other Names: Dynamic arterial elastance
  Arms: administration of norepinephrine by dynamic elastance
Drug: Norepinephrine — The usual procedure of withdrawal norepinephrine is based on hemodynamic parameters (blood pressure, cardiac output), clinical (cutaneous perfusion, mottling, hourly diuresis) and biological (SVO2, arterial lactate).
  Other Names: Control
  Arms: control administration of norepinephrine

SUMMARY:
After cardiac surgery, vasoplegic syndrome is a hemodynamic state characterized by profound hypotension associated with a decrease in systemic vascular resistance. The care of this disease is based on the intravenous administration of a vasopressor, usually norepinephrine. During the recovery phase, weaning of norepinephrine, is an important step in which any lack of preload (blood volume) initial or secondary can be, and increase tissue malperfusion.

ELIGIBILITY:
Inclusion Criteria:

* Major patient ≥ 18 years
* Patient operated a cardiac surgery for myocardial revascularization (CABG surgery) or surgical correction of valvular or combined surgery (CABG and valve disease) or surgery the ascending aorta and cardiac surgery with vasoplegic syndrome treated by norepinephrine
* Signed consent
* Affiliation to social assurance

Exclusion Criteria:

* Permanent atrial fibrillation
* Treatment with dobutamine and/or epinephrine
* Pregnant woman
* Patient under guardianship or private public law
* Internal pacemaker
* Hypothermia
* Patient refusal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The duration of treatment with norepinephrine. | Day 28
  Mean duration time of norepinephrine administration calculated in hours

SECONDARY OUTCOMES:
The total dose of norepinephrine infused during the study period | Day 28
ICU duration of stay in day | Day 28
Total urine output in ml during the study period | Day 28
Total of crystalloid an colloid infused during the study period (ml) | Day 28
the rate of arterial lactate at the end of norepinephrine administration | Day 28
Incidence of postoperative atrial arrhythmias (Ac/Fa, Ventricular tachycardia, Ventricular flutter, Ventricular fibrillation) during the study period | Day 28
SOFA score | Day 28
  SOFA score measured at the end of norepinephrine administration

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Grégoire Guinot, Doctor, Principal Investigator — CHU Amiens-Picardie
Locations (1):
- CHU Amiens-Picardie, Amiens, Picardie, France

REFERENCES:
- [Background] Guinot PG, Bernard E, Levrard M, Dupont H, Lorne E. Dynamic arterial elastance predicts mean arterial pressure decrease associated with decreasing norepinephrine dosage in septic shock. Crit Care. 2015 Jan 19;19(1):14. doi: 10.1186/s13054-014-0732-5. PMID 25598221
- [Result] Guinot PG, Abou-Arab O, Guilbart M, Bar S, Zogheib E, Daher M, Besserve P, Nader J, Caus T, Kamel S, Dupont H, Lorne E. Monitoring dynamic arterial elastance as a means of decreasing the duration of norepinephrine treatment in vasoplegic syndrome following cardiac surgery: a prospective, randomized trial. Intensive Care Med. 2017 May;43(5):643-651. doi: 10.1007/s00134-016-4666-z. Epub 2017 Jan 24. PMID 28120005